CLINICAL TRIAL: NCT02272062
Title: Patient-Reported Preferences Affecting Revascularization Decisions
Acronym: PREPARED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00055866
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Coronary Artery Disease; Angina Pectoris
Keywords: Coronary artery disease; Angina; Shared decision-making; Patient preferences; Percutaneous coronary intervention; Coronary artery bypass graft
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Patient Preference

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preferences Not Provided (No Intervention): Subjects will complete a shared decision-making tool and express preferences regarding treatment for coronary artery disease, but these preferences will NOT be shared with the treating clinicians.
- Preferences Provided (Experimental): Subjects will complete a shared decision-making tool and express preferences regarding treatment for coronary artery disease, and these preferences WILL be shared with the treating clinicians.
  Interventions: Other: Decision-making tool for coronary artery disease treatment

INTERVENTIONS:
Other: Decision-making tool for coronary artery disease treatment — A brief internet-based tool will provide education about coronary artery disease and assess patient preferences regarding treatment options (medical management, percutaneous coronary intervention, or coronary artery bypass graft). This information will be provided to the treating interventional cardiologist at the time of coronary angiography in the treatment group.
  Arms: Preferences Provided

SUMMARY:
Selection of a treatment strategy for patients with symptoms due to coronary artery disease requires consideration of patient preferences. In current clinical practice, patient preferences for treatment may not be known prior to diagnostic coronary angiography. The investigators will test an internet-based shared decision-making tool which will provide education and solicit preference information prior to angiography. The investigators seek to determine if this tool can accurately assess patient preferences, and if these preferences will lead to a change in clinical management.

DETAILED DESCRIPTION:
Selecting a treatment strategy for patients with symptomatic coronary artery disease (CAD) requires integrated consideration of symptom burden, patient preferences, and practice guidelines. In many clinical scenarios, there is equipoise regarding the need to revascularize (percutaneous coronary intervention (PCI) vs. medical management) and/or the type of revascularization (PCI vs. bypass surgery). Patients may have minimal direct input in the decision to proceed to a revascularization procedure, especially in the case of ad hoc PCI.

There is little guidance in the literature regarding strategies to improve patient participation in revascularization decisions. There is no shared decision-making tool to provide accessible information to the interventional cardiologist prior to PCI. An educational program that provides basic information regarding CAD and revascularization procedures could lead to improved patient knowledge and informed participation in these critical decisions. A clinical survey that assesses patient symptom burden and preferences could provide valuable information to physicians at the time of angiography. The investigators aim to test a clinical tool that addresses both of these needs and can be administered in the pre-procedure area immediately prior to angiography. If successful, this tool could lead to greater informed patient participation in revascularization procedures and improved patient satisfaction.

First, the investigators will conduct a pre-post analysis. The first 100 enrolled patients will undergo usual care without the use of the decision-making tool. Surveys prior to angiography and at 3 months will test knowledge and decisional self-efficacy. Subsequently, 200 patients will utilize the decision-making tool and will complete the same surveys. Comparison of these groups will test the ability of the decision-making tool to improve knowledge about CAD and accurately assess preferences.

Among the 200 patients utilizing the decision-making tool, patients will be randomly assigned to have, or not have, their preferences shared with the interventional cardiologist at the time of catheterization. This randomized portion of the study will test the impact of patient preferences on treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to the catheterization laboratory for diagnostic coronary angiography with a reasonable expectation of coronary artery disease, defined as chronic stable angina, chest pain with a positive functional study, unstable angina, or non-ST segment elevation myocardial infarction.

Exclusion Criteria:

* Unable to provide informed consent
* Unable to speak or read English
* Critical illness
* When a delay in angiography to administer the decision aid could lead to adverse clinical outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Concordance of patient preference with delivered treatment | 3 months
  Among patients with significant coronary artery disease on diagnostic angiography, the percentage of subjects with delivered therapy (medical management, percutaneous coronary intervention, coronary artery bypass graft) identical to preferences expressed prior to angiography.

SECONDARY OUTCOMES:
Knowledge | Within 2 hours of angiography
  Performance on a 6-item knowledge questionnaire
Knowledge | 3 months
  Performance on a 6-item knowledge questionnaire
Decisional conflict | Within 2 hours of angiography
  Performance on a 16-item scale assessing decisional self-efficacy
Patient satisfaction | Within 2 hours of angiography
  Performance on the decisional regret scale
Patient satisfaction | 3 months
  Performance on the decisional regret scale
Informed values congruence | Within 2 hours of angiography
  Concordance of the subject's stated preference for treatment with treatment-specific results from the Patient Preferences Questionnaire for Angina Treatment
Angina | 3 months
  7-item Seattle Angina Questionnaire
Ad hoc percutaneous coronary intervention | 3 months
  Percentage of percutaneous coronary intervention performed at time of diagnostic angiography

CONTACTS AND LOCATIONS:
Overall Officials: Manesh Patel, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

REFERENCES:
- [Derived] Doll JA, Jones WS, Lokhnygina Y, Culpepper S, Parks RL, Calhoun C, Au DH, Patel MR. PREPARED Study: A Study of Shared Decision-Making for Coronary Artery Disease. Circ Cardiovasc Qual Outcomes. 2019 Feb;12(2):e005244. doi: 10.1161/CIRCOUTCOMES.118.005244. PMID 30764651